CLINICAL TRIAL: NCT03538028
Title: A Phase 1 Open-Label, Dose-Escalation, Safety and Tolerability Study of INCAGN02385 in Participants With Select Advanced Malignancies
Brief Title: A Safety and Tolerability Study of INCAGN02385 in Select Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 2385-101
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Cervical Cancer; Microsatellite Instability (MSI)-High Endometrial Cancer; Gastric Cancer (Including Stomach and Gastroesophageal Junction [GEJ]); Esophageal Cancer; Hepatocellular Carcinoma; Melanoma (Uveal Melanoma Excluded); Merkel Cell Carcinoma; Mesothelioma; MSI-high Colorectal Cancer; Non-small Cell Lung Cancer (NSCLC); Ovarian Cancer; Squamous Cell Carcinoma of the Head and Neck (SCCHN); Small Cell Lung Cancer (SCLC); Renal Cell Carcinoma (RCC); Triple-negative Breast Cancer; Urothelial Carcinoma; Diffuse Large B-cell Lymphoma
Keywords: lymphocyte activation gene (LAG); LAG-3; advanced solid tumor; metastatic solid tumor; relapsed/refractory DLCBL
MeSH Terms: conditions — Uterine Cervical Neoplasms; Microsatellite Instability; Stomach Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Merkel Cell; Mesothelioma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCAGN02385 (Experimental): Part 1: INCAGN02385 at the protocol-defined starting dose administered every 2 weeks (Q2W), with dose escalation to determine the maximum tolerated dose or pharmacologically active dose. Part 2: INCAGN02385 administered Q2W or Q4W at the recommended dose(s) from Part 1.
  Interventions: Biological: INCAGN02385

INTERVENTIONS:
Biological: INCAGN02385 — INCAGN02385 administered as an intravenous infusion over 30 minutes.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and preliminary efficacy of INCAGN02385 in participants with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Disease progression after treatment with available therapies that are known to confer clinical benefit, or intolerant to treatment, or refuse noncurative standard treatment. There is no limit to the number of prior treatment regimens.
* Participants with advanced or metastatic cervical cancer, MSI-high endometrial cancer, gastric cancer (including stomach and GEJ), esophageal cancer, hepatocellular carcinoma, melanoma (uveal melanoma excluded), Merkel cell carcinoma, mesothelioma, MSI-high colorectal cancer, NSCLC, ovarian cancer, SCCHN, SCLC, RCC, triple-negative breast cancer, and urothelial carcinoma, or alternative immunogenic tumor types with medical monitor approval. Participants with DLBCL may participate in Part 2 of the study.
* Presence of measureable disease based on RECIST v1.1 for solid tumors or the Lugano classification for DLBCL.
* Willingness and ability to safely undergo pretreatment and on-treatment tumor biopsies.
* Eastern Cooperative Oncology Group performance status 0 or 1.

Exclusion Criteria:

* Laboratory and medical history parameters outside the protocol-defined range.
* Transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 14 days before study Day 1.
* Receipt of anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Receipt of a live vaccine within 30 days of planned start of study drug.
* Active autoimmune disease that required systemic treatment in the past.
* Known active CNS metastases and/or carcinomatous meningitis.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry. See protocol-defined exceptions.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* Active infection requiring systemic therapy.
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.
* Known history of HIV (HIV 1/2 antibodies).
* Prior treatment with an anti-LAG-3 antibody for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | Up to 12 months
  TEAE defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Cmax of INCAGN02385 | Up to 12 months
  Maximum observed plasma concentration.
Tmax of INCAGN02385 | Up to 12 months
  Time to maximum plasma concentration.
Cmin of INCAGN02385 | Up to 12 months
  Minimum observed plasma concentration during the dosing interval.
AUC0-t of INCAGN02385 | Up to 12 months
  Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration.
Objective response rate (ORR) in participants with advanced or metastatic solid tumors | Up to 12 months
  Defined as the percentage of participants having complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Disease control rate (DCR) in participants with advanced or metastatic solid tumors | Up to 12 months
  Defined as percentage of participants having CR, PR, or stable disease (SD) as best on-study response.
Duration of response (DOR) in participants with advanced or metastatic solid tumors | Up to 12 months
  Defined as the time from earliest date of disease response (CR or PR) until earliest date of disease progression per RECIST v1.1 or death from any cause, if occurring sooner than progression.
Progression-free survival (PFS) in participants with advanced or metastatic solid tumors | Up to 12 months
  Defined as the time from date of first dose of study drug until the earliest date of disease progression per RECIST v1.1 or death from any cause if occurring sooner than progression.
ORR in participants with diffuse large B-cell lymphoma (DLBCL) | Up to 12 months
  Defined as the percentage of participants with a CR/complete metabolic response (CMR) or PR/partial metabolic response (PMR) per the Lugano Classification.
DOR in participants with DLBCL | Up to 12 months
  Defined as the time from first documented evidence of CR/CMR or PR/PMR until disease progression per radiographic disease assessment or death from any cause among participants who achieve an objective response.
PFS in participants with DLBCL | Up to 12 months
  Defined as the time from the date of the first dose of study drug until the earliest date of disease progression per radiographic disease assessment or death from any cause if occurring sooner than progression.

CONTACTS AND LOCATIONS:
Overall Officials: John Janik, MD, Study Director — Incyte Corporation
Locations (4):
- United States (4):
  - The Angeles Clinic and Research Center, Los Angeles, California
  - Hackensack Medical Center, Hackensack, New Jersey
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No